CLINICAL TRIAL: NCT04608903
Title: Salutary Effects of Sulforaphane for Patients With Chronic Kidney Disease
Brief Title: Effects of Sulforaphane for Patients With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: DeniseMafra11
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Sulforaphane group or Placebo group. Thus, 52 participants with CKD under conservative treatment will be recruited at the Renal Nutrition Clinic of UFF and 70 patients under regular HD treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulforaphane Group (Experimental): Administration of 4g L-sulforaphane per day, for 2 months and after the washout period (2 months) the groups will be crossed and will receive the same amount of placebo as the other group for 2 months.
  Interventions: Dietary Supplement: L-sulforaphane 1%
- Placebo Group (Placebo Comparator): Administration of 4g of corn starch colored with chlorophyll, per day, for 2 months and then after the washout period (2 months) the groups will be crossed and will receive the same amount of sulfarophane as the treatment group.
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: L-sulforaphane 1% — Administration of 4g L-sulforaphane per day, for 2 months
  Arms: Sulforaphane Group
Dietary Supplement: Placebo Group — Administration of 4g corn starch colored with chlorophyll, per day, for 2 months
  Arms: Placebo Group

SUMMARY:
Patients with Chronic Kidney Disease (CKD) have many complications associated with inflammation, oxidative stress and intestinal dysbiosis, which are closely related to the progression of kidney failure and cardiovascular disease. Sulforaphane, an isothiocyanate found in cruciferous vegetables (Family: Brassicaceae) is recognized as one of the most important activators of erythroid nuclear factor 2 related to factor 2 (Nrf2). However, clinical evidence to assess the effects of sulforaphane in patients with CKD is scarce, and there are no studies that have investigated its effects on the expression of genes and markers related to inflammation in these patients. Thus, the present project proposes a longitudinal study of the clinical trial type that aims to evaluate the effects of sulforaphane on transcription factors and inflammatory markers in patients with CKD.

DETAILED DESCRIPTION:
This is a longitudinal, randomized, crossover study with patients with CKD on hemodialysis and in non-dialysis patients.

Both groups will receive 4g of sulforaphane per day for 2 months and the placebo group will receive 4g of corn starch colored with chlorophyll for 2 months. Peripheral blood mononuclear cells (PBMC) are being isolated for expression of Nrf2, NF-kB, and NADPH quinone oxidoreductase 1 (NQO1), HO-1, VCAM-1, E-selectin, NLRP3, IL-1B, IL 18, PGC1-α, sentrins, NRF2, NRF-1 e TFAM mRNA expression by a quantitative real-time polymerase chain reaction. Antioxidant enzymes activity (catalase-CAT and glutathione peroxidase-GPx), high-sensitivity C-reactive protein (hs-CRP) will be assessed using an enzyme-linked immunosorbent assay (ELISA).The serum concentration of other cytokines and growth factors will be detected by means of a multiparametric immunoassay based on magnetic microspheres marked with XMap (Luminex Corp, USA) before and after supplementation.

ELIGIBILITY:
Criteria

Inclusion Criteria:

* Aged 18 to 75 years
* Clinical diagnosis of Chronic Kidney Disease
* Conservative treatment group: CKD stages 3 and 5 receiving nutritional treatment for at least 6 months
* Hemodialysis group: Hemodialysis patients for more than 6 months

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Autoimmune diseases
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Antioxidant and anti-inflammatory biomarker | 6 months
  Get blood samples to evaluate the supplementation effects in antioxidant and anti-inflammatory biomarker- nuclear receptor factor 2 (Nrf2)
Inflammatory biomarker | 6 months
  Get blood samples to evaluate the supplementation effects in inflammatory biomarker- factor nuclear kappa B (NFkB)

SECONDARY OUTCOMES:
Uremic toxins | 6 months
  Get blood samples to evaluate the supplementation effects on uremic toxins plasma levels

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardozo LFMF, Alvarenga LA, Ribeiro M, Dai L, Shiels PG, Stenvinkel P, Lindholm B, Mafra D. Cruciferous vegetables: rationale for exploring potential salutary effects of sulforaphane-rich foods in patients with chronic kidney disease. Nutr Rev. 2021 Oct 11;79(11):1204-1224. doi: 10.1093/nutrit/nuaa129. PMID 33338213